CLINICAL TRIAL: NCT03554382
Title: PERson-centredness in Hypertension Management Using Information Technology (PERHIT) Study
Brief Title: Efficient Self-management of Chronic Disease Using Health Information Technology - a Study on Hypertension
Acronym: PERHIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: the Kamprad Family Foundation (Unknown); Swedish Heart Lung Foundation (Other); Clinical Studies Sweden - Forum South (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERHIT
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; High Blood Pressure
Keywords: person-centred care (PCC); self-efficacy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomization to study groups occurs after completion of informed consent, baseline assessments and questionnaires. Patients are randomly assigned in a 1:1 ratio to either the intervention group or the control group. The CONSORT-EHEALTH checklist will be followed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Daily use of interactive mobile phone-based system to support self-management of hypertension: a) relevant items on drug side effects related to patient's drug regimen; and b) blood pressure.
  Interventions: Other: system to support self-management of hypertension
- Control (No Intervention): No study intervention will be made in the control group; they will receive "treatment as usual".

INTERVENTIONS:
Other: system to support self-management of hypertension — The patients are provided with a home BP monitor. Thereafter they will be asked to use the self-management support system and self-report, once daily in the evening, via their own mobile phone during eight weeks. At each occasion, the patients first answer the questions on wellbeing, symptoms, lifestyle, medication intake and side effects and then measure their BP and pulse, and when these data (mean of three readings) are input into the mobile phone, they automatically register in the database. During intervention the paient has regular access to self-reported data via graphs
  Arms: intervention

SUMMARY:
Background:

Hypertension is an increasing global problem and measures are needed against the emerging hypertensive burden. Management of the risk factor hypertension consists of medical treatment in conjunction with lifestyle adjustment, whereby lifestyle adjustment is the preventive cornerstone but has also been proven to contribute to BP reduction among those already receiving medical drug treatments. Non-adherence is a significant barrier to successful hypertension management.

Goal:

To improve management of hypertension in daily life from a person-centred perspective, utilizing information and communication technology, and further to decrease complications of hypertension. To increase the proportion of persons with hypertension obtaining a BP goal =<140/90 mmHg and to conduct a health economic evaluation of our intervention.

Plan:

The investigators will conduct a multi-centre randomized controlled trial in 36 primary care centres in three counties in Sweden. There will be approximaely 430 patients in each group. BP will be measured in a standardized manner, laboratory tests taken and questionnaires answered at baseline, after eight weeks and after a year in both the intervention and the control group. Register data on health care resource one year before baseline and for the full study period will be retrieved for participants in both study groups.

Singificance:

The intervention is expected to improve adherence to treatment and a significant lowering of the blood pressure. Hospitalization rates are lower among persons with hypertension that adheres to their medication. By improving treatment of hypertension the hope is to decrease complications and morbidity due to hypertension and thereby hospitalization and health care costs. Due to the generic nature of the technology involved, the self-management system can easily be adapted to monitor other chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of hypertension
* On treatment with at least one antihypertensive drug
* Understanding of Swedish in order to be able to provide informed consent and to make use of the mobile phone based self-management support system.
* Mobile phone (patients will use their own mobile, but have the possibility to borrow one if needed)
* Patient at a primary healthcare centre in any of four participating healthcare regions in Sweden (Skåne, Västra Götaland, Östergötland, and Jönköping)

Exclusion Criteria:

* Secondary hypertension
* Terminal illness
* Pregnancy-induced hypertension
* Cognitive impairment
* Impaired vision (not able to read messages on mobile phone)
* Psychotic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 971 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | 12 months
  mean of three BP Readings at each timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Midlöv, MD, Principal Investigator — Lund University
Locations (4):
- Sweden (4):
  - Solklart vård i Bjuv, Bjuv
  - Wetterhälsan, Jönköping
  - Vårdcentralen Kärna, Linköping
  - Adina Hälsans Vårdcentral Nol, Nol

REFERENCES:
- [Derived] Ekholm M, Andersson U, Nilsson PM, Kjellgren K, Midlov P. Evaluation of self-monitoring of blood pressure in the PERHIT study and the impact on glomerular function. Blood Press. 2024 Dec;33(1):2399565. doi: 10.1080/08037051.2024.2399565. Epub 2024 Sep 9. PMID 39250514
- [Derived] Vestala H, Bendtsen M, Midlov P, Kjellgren K, Eldh AC. Is patient participation in hypertension care based on patients' preferences? A cross-sectional study in primary healthcare. Eur J Cardiovasc Nurs. 2024 Dec 16;23(8):903-911. doi: 10.1093/eurjcn/zvae085. PMID 38805264
- [Derived] Andersson U, Nilsson PM, Kjellgren K, Harris K, Chalmers J, Ekholm M, Midlov P. Variability in home blood pressure and its association with renal function and pulse pressure in patients with treated hypertension in primary care. J Hum Hypertens. 2024 Mar;38(3):212-220. doi: 10.1038/s41371-023-00874-2. Epub 2023 Nov 15. PMID 37968455
- [Derived] Andersson U, Nilsson PM, Kjellgren K, Hoffmann M, Wennersten A, Midlov P. PERson-centredness in Hypertension management using Information Technology: a randomized controlled trial in primary care. J Hypertens. 2023 Feb 1;41(2):246-253. doi: 10.1097/HJH.0000000000003322. Epub 2022 Nov 18. PMID 36394295
- [Derived] Andersson U, Bengtsson U, Ranerup A, Midlov P, Kjellgren K. Patients and Professionals as Partners in Hypertension Care: Qualitative Substudy of a Randomized Controlled Trial Using an Interactive Web-Based System Via Mobile Phone. J Med Internet Res. 2021 Jun 3;23(6):e26143. doi: 10.2196/26143. PMID 34081021